CLINICAL TRIAL: NCT01536925
Title: Biobehavioral Studies of Opioid Seeking Behavior: Yohimbine and Hydrocortisone Effects
Brief Title: Studies of Opioid Seeking Behavior: Yohimbine and Hydrocortisone Effects
Acronym: YHO
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Professor, Wayne State University
Other Study IDs: YHO-1; R01DA015462-06A1 (NIH)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Heroin Dependence; Opioid-Related Disorders
Keywords: Behavioral Economics; Drug self administration; Opioid
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This research deals with behaviors that are part of opioid dependence. The purpose is to study the extent to which stress and other factors, including money and amount of work effort, affect opioid choice. Specifically, the investigators will examine the effects of three issues/factors. The first is how hard participants are willing to work to obtain an opioid drug; the second is how much opioid drug would participants choose instead of money; and the third factor is how much participant's opioid drug choices are influenced after they are administered the drugs yohimbine and hydrocortisone, both of which could produce stress-like symptoms.

DETAILED DESCRIPTION:
Phase 1: Participants will first be an outpatient and must come to the Tolan Park Medical Building daily to receive buprenorphine doses. This phase will last at least 10 days or longer. Three times per week during the first two weeks (i.e., on 6 different days), participants will be asked to provide urine samples and to complete questionnaires that ask about opiate withdrawal symptoms.

Phase 2: Participants will then live on an inpatient research unit (located in Detroit Michigan) for at least 16 consecutive nights and possibly up to 18 consecutive nights. Participants will continue on the same dose of buprenorphine as in phase 1.

During this stay they will participate in a total of 11 experimental sessions. Participants will take part in multiple trials in which they have the opportunity to choose drug, hydromorphone, or money. Hydromorphone is a heroin-like opioid. During the first two test sessions, participants will receive a sample of the drug doses that can be chosen. Before each of the final 9 test sessions begin, participants will be given a capsule containing either different doses of the drug yohimbine or a placebo (blank). Yohimbine is a drug that has been shown to produce a "stress"-like response in humans. Then participants will be given a capsule that contains either different doses of the drug hydrocortisone or a placebo (blank). Hydrocortisone is also a drug that can produce a "stress"-like response in humans. Then participants will have the opportunity to choose either drug or money by using a computer to earn choices. Respiration rate, oxygen saturation, heart rate, and blood pressure will be monitored throughout choice trials. Self-report questionnaires will be completed at different times during the study.

Phase 3: After participants have completed the experimental procedures, they will again come to the Tolan Park Medical Building daily to receive buprenorphine doses. The dose of buprenorphine will be gradually decreased so that they will eventually be free from medication. This will take three weeks. We will administer questionnaires and collect urine samples three times each week.

ELIGIBILITY:
Inclusion Criteria:

* Opioid dependent, as determined by structured clinical interview for DSM-IV (SCID) and Addiction Severity Index (ASI)
* Positive urine test for opiates
* Willing to use an adequate form of contraception for the duration of the study.
* Reads and writes English
* Participants must be in generally good health to be eligible. All candidates will receive a routine medical exam (history and physical) with standard laboratory tests (including blood and urine samples, EKG, mandatory TB testing, and voluntary HIV testing).

Exclusion Criteria:

* No candidate who has a current DSM-IV Axis I disorder other than Drug Dependence or a history of serious psychiatric problems (e.g. psychosis, bipolar or major depression) will be allowed to participate.
* Candidates meeting criteria for opioid or nicotine dependence will not be excluded, but those with other Substance Dependence disorders will be excluded. Those with Abuse of Alcohol, Cannabis, Cocaine, or Benzodiazepines will not be excluded, but participants must provide an alcohol free breath specimen, and a benzodiazepine free urine sample.
* No candidate with medical (neurological, cardiovascular, pulmonary or systemic) disorders will be allowed to participate. This will be determined with history and physical exam, standard laboratory testing (blood and urine), EKG, and TB tests (to avoid transmitting this communicable disease on the residential unit or in the laboratory).
* Candidates with evidence of cognitive impairment (based on reading ability and comprehension, will be excluded.
* Female candidates who are pregnant (urine pregnancy test), lactating, or not using adequate birth control methods (self-report) will be excluded.
* Candidates with injection phobia, or seeking treatment for opioid dependence will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Heroin dependent research volunteers
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-12; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Derived] Stoltman JJ, Woodcock EA, Lister JJ, Greenwald MK, Lundahl LH. Exploration of the telescoping effect among not-in-treatment, intensive heroin-using research volunteers. Drug Alcohol Depend. 2015 Mar 1;148:217-20. doi: 10.1016/j.drugalcdep.2015.01.010. Epub 2015 Jan 19. PMID 25630964